CLINICAL TRIAL: NCT02089178
Title: Comparison of the Effect of Total Intravenous Anesthesia and Inhalation Anesthesia on Cancer Cell Cytotoxicity, Micrometastasis and Recurrence of Tumor in Patients Undergoing Breast Tumor Resection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study costed more than expected, so the investigators decided to end it.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2013-0937
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: total intravenous anesthesia, inhalation anesthesia, cancer cell cytotoxicity, breast tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, Intravenous; Anesthesia, Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous (Experimental): the total intravenous anesthesia group
  Interventions: Procedure: intravenous anesthesia; Drug: propofol-remifentanil
- inhalation (Active Comparator): the inhalation anesthesia group
  Interventions: Procedure: inhalation anesthesia; Drug: sevoflurane-remifentanil

INTERVENTIONS:
Procedure: intravenous anesthesia — total intravenous anesthesia group: propofol-remifentanil
  Arms: intravenous
Procedure: inhalation anesthesia — inhalation anesthesia group: sevoflurane-remifentanil
  Arms: inhalation
Drug: propofol-remifentanil
  Arms: intravenous
Drug: sevoflurane-remifentanil
  Arms: inhalation

SUMMARY:
The purpose of this study is to compare the effect of total intravenous anesthesia and inhalation anesthesia on cancer cell cytotoxicity, micrometastasis and recurrence of tumor in patients undergoing breast tumor resection. Using propofol-remifentanil in total intravenous anesthesia group and sevoflurane -remifentanil in inhalation anesthesia group.

ELIGIBILITY:
Inclusion Criteria:

* patient between 20 and 65 of age with ASA physical status Ⅰ-Ⅲ
* breast cancer patients with no sign of local invasion (adjacent organs) and distant metastasis revealed by imaging studies
* surgery performed by the same surgical team

Exclusion Criteria:

* ASA physical status Ⅳ
* hepatic and renal impairment
* diabetes or other endocrine disorders
* body mass index > 35 kg/m2
* immune disorders or immunosuppressive therapy
* steroid treatment in the last 6 months
* inflammation

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
number of NK cell | at 24 hour after surgery.
  comparison of the effect of total intravenous anesthesia and inhalation anesthesia on cancer cell cytotoxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea